CLINICAL TRIAL: NCT01419626
Title: Antiplaque and Antigingivitis Efficacy of Interdental Cleaning Using an Experimental Device in Combination With an Essential-oil Containing Mouthrinse
Brief Title: A Study to Determine the Effects of Adding an Experimental Device With Mouthrinse to Oral Care Regimen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UNKPLT0008
Record Dates: First submitted 2011-08-17; First posted 2011-08-18 (Estimated); Results first posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-11

CONDITIONS: Gingivitis
Keywords: Dental Plaque; Interdental Cleaning Device
MeSH Terms: conditions — Gingivitis; Dental Plaque | interventions — Hydrotherapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Negative Control (No Intervention): Subjects will be instructed to follow their usual oral hygiene habits with the provided toothbrush and toothpaste.
- Device with Water (Sham Comparator): Subjects will be instructed to follow their usual oral hygiene habits with the provided toothbrush and toothpaste, and to use their assigned product once a day for a period of 4 weeks.
  Interventions: Device: Interdental cleaning device with water
- Device with Mouthrinse (Experimental): Subjects will be instructed to follow their usual oral hygiene habits with the provided toothbrush and toothpaste, and to use their assigned product once a day for a period of 4 weeks.
  Interventions: Device: Interdental cleaning device with essential-oil mouthrinse

INTERVENTIONS:
Device: Interdental cleaning device with water — Subjects will be instructed to follow their usual oral hygiene habits with the provided toothbrush and toothpaste, and to use their assigned product once a day for a period of 4 weeks.
  Other Names: Regulation # 872.6510 with water
  Arms: Device with Water
Device: Interdental cleaning device with essential-oil mouthrinse — Subjects will be instructed to follow their usual oral hygiene habits with the provided toothbrush and toothpaste, and to use their assigned product once a day for a period of 4 weeks.
  Other Names: Regulation # 872.6510 with Mouthrinse # 19292-116A
  Arms: Device with Mouthrinse

SUMMARY:
The study will determine the effects of adding mechanical plaque control to a person's oral care regimen. Participants who qualify to participate in the study will will have an equal chance of being assigned to one of three groups. They will be asked to follow their assigned oral care regimen, fill out subject diaries as instructed, and return to the clinic two weeks and four weeks afterward to have their mouths examined.

DETAILED DESCRIPTION:
At baseline, the prescreened subjects will present to the clinical site for baseline examinations (oral exam, plaque, gingivitis and gingival bleeding assessments) having refrained from oral hygiene for at least 12 hours, but no more than 18 hours and from eating for at least 2 hours prior to that examination. After the baseline oral examinations, and assessment of other inclusion/exclusion criteria, qualifying subjects will be randomly assigned to one of the three treatment groups. Immediately following this randomization, all subjects will begin their regimen of brushing with a manual toothbrush while two of the groups will also receive an experimental interdental cleaning device to use either with water or with an assigned mouthrinse following the label instructions described on the experimental device label. Subjects who are assigned to the negative control group will use the manual toothbrush and provided toothpaste as their sole mean of oral hygiene. Subjects assigned to the Device-only control group will brush with a manual toothbrush and use the Experimental Interdental Cleaning Device with water. Finally, those subjects randomized to the test group will brush with a manual toothbrush and use the experimental interdental cleaning device in combination with a marketed antiseptic mouthrinse.

Subjects will brush twice-a-day and if assigned, will use the experimental interdental cleaning device once-a-day for 4 weeks, post-brushing, according to instructions given by the study personnel. The first oral hygiene procedure will be conducted under supervision of study personnel at the research site. All other study material usage will be unsupervised and the subjects will be required to maintain a Diary Card to document daily oral hygiene routine. Compliance will be evaluated at each visit by reviewing the subject diaries and, when applicable, by weighing residual volumes of returned mouthrinse.

Subjects will refrain from the use of any interdental cleaning device, unless assigned by the randomization schedule (i.e., not to use dental floss, toothpick, etc), unless it is used to remove impacted food between the teeth, during the course of the study. No other oral hygiene procedures will be permitted, including teeth cleaning or dental work except for an emergency.

At the two and four-week visits, the Modified Gingival Index (MGI), the Bleeding Index (BI) and the Turesky modification of the Quigley-Hein Plaque Index (PI) will be scored and the oral tissue examinations performed. At the two and four-week visits, subjects will not have used their test materials for at least 12 hours, but no more than 18 hours.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and follow the requirements of the study (including availability on scheduled visit dates) based upon research site personnel's assessment.
* Able to provide written informed consent; volunteers must read, sign, and receive a copy of the signed Informed Consent Form after the nature of the study has been fully explained.
* Males and females 18 years of age or older, in good general and oral health, except gingivitis.
* A minimum of 20 natural teeth with scorable facial and lingual surfaces. Teeth that are grossly carious, extensively restored, orthodontically banded, abutments, exhibiting severe generalized cervical and/or enamel abrasion, or third molars will not be included in the tooth count.
* A gingival index ≥ 1.75 according to the Modified Gingival Index.
* A plaque index ≥ 1.95 according to the Turesky modification of the Quigley-Hein Plaque Index scored on six surfaces per tooth.
* Gingival Bleeding Index ≥ 0.1.
* Absence of significant oral soft tissue pathology, excluding plaque-induced gingivitis, based on a visual examination and at the discretion of the Investigator.
* Absence of moderate/advanced periodontitis based on a clinical examination (ADA Type III, IV).
* Absence of fixed or removable orthodontic appliance or removable partial dentures.
* Are willing and able to fully understand and comply with the written and verbal study instructions provided in English
* Agree to return all study materials at the final visit (week 4).

Exclusion Criteria:

* History of significant adverse effects, including sensitivities or suspected allergies, following use of oral hygiene products such as toothpastes and mouthrinses and red food dye.
* History of serious medical conditions that, at the discretion of the Investigator, will disqualify the subject, such as having have a cardiac pacemaker or AICD.
* History of rheumatic fever, heart murmur, mitral valve prolapse or other conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures.
* Antibiotic, anti-inflammatory or anticoagulant therapy during the study or within the 2 weeks prior to the baseline exam.
* Regular use of chemotherapeutic antiplaque/antigingivitis products such as triclosan, essential oil, cetylpyridinium chloride, or chlorhexidine containing mouthrinses within the 2 weeks prior to baseline.
* Current or history of alcohol or drug abuse, and those who smoke more than one pack of cigarettes per day
* Females who are pregnant or breastfeeding.
* Known sensitivity to the investigational product.
* Significant unstable or uncontrolled medical condition which may interfere with a subject's participation in the study.
* Participation in any clinical study within 30 days of Visit 1.
* Relative, partner or staff of any clinical research site personnel.
* A member of the same household (i.e. residing in the same house) is a participant in this study.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* Are employed by an oral healthcare products company or dental research institution (i.e., dental school: administrative staff, assistants, hygienists, and research students).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-07-31 (Actual); Primary Completion 2011-08-31 (Actual); Study Completion 2011-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo WB Araujo, DDS,MS,PhD, Study Director — Johnson & Johnson Consumer and Personal Products Worldwide
Locations (1):
- BioSci Research America, Inc, Las Vegas, Nevada, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Negative Control Group (Toothbrushing Only): Following randomization, participants started brushing teeth with a manual toothbrush (Advanced Design Toothbrush - ADR # PR-000172) twice daily with provided toothpaste as their sole means of oral hygiene for up to 4 Weeks.
- Device Control Group (Toothbrushing, Device + Water): Following randomization, participants started brushing teeth with a manual toothbrush (Advanced Design Toothbrush - ADR # PR-000172) and provided toothpaste twice daily with an experimental interdental cleaning device to use with water once a day after brushing for up to 4 Weeks.
- Test Group (Toothbrushing, Device+ Oil-containing Mouthrinse): Following randomization, participants started brushing teeth with a manual toothbrush (Advanced Design Toothbrush - ADR # PR-000172) provided toothpaste twice daily with an experimental interdental cleaning device to use with the assigned marketed antiseptic mouthrinse (essential oil-containing mouthrinse) once a day after brushing for up to 4 Weeks.
Period: Overall Study
Arm/Group | Negative Control Group (Toothbrushing Only) | Device Control Group (Toothbrushing, Device + Water) | Test Group (Toothbrushing, Device+ Oil-containing Mouthrinse)
Started | 46 | 47 | 47
Completed | 42 | 44 | 44
Not Completed | 4 | 3 | 3
Not completed — Protocol Violation | 3 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Negative Control Group (Toothbrushing Only) | Device Control Group (Toothbrushing, Device + Water) | Test Group (Toothbrushing, Device+ Oil-containing Mouthrinse) | Total
Number analyzed (Participants) | 46 | 47 | 47 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (12.26) | 34.5 (11.27) | 34.9 (10.35) | 35.6 (11.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 38 | 26 | 90
  Male | 20 | 9 | 21 | 50
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46 | 47 | 47 | 140

OUTCOME MEASURES:

1. Primary Outcome: Interproximal Mean Plaque Index at Week 4
Description: Plaque area was scored using the Turesky modification of the Quigley-Hein Plaque Index (PI), on six surfaces (distobuccal, midbuccal and mesiobuccal, distolingual, midlingual and mesiolingual) of all scorable teeth, using following score range; 0: indicates no plaque; 1: separate flecks or discontinuous band of plaque on the gingival (cervical) margin; 2: thin (up to 1 millimeter [mm]), continuous band of plaque at the gingival margin; 3: band of plaque wider than 1mm but less than1/3 of the surface; 4: plaque covering 1/3 or more, but less than 2/3 of the surface; 5 plaque covering 2/3 or more of the surface.
Time Frame: Week 4
Population: Full analysis set (FAS) included all randomized participants who used study product and had baseline and at least one data for mean PI post baseline.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Test Group (Toothbrushing, Device + Oil-containing Mouthrinse): Following randomization, participants started brushing teeth with a manual toothbrush (Advanced Design Toothbrush - ADR # PR-000172) provided toothpaste twice daily with an experimental interdental cleaning device to use with the assigned marketed antiseptic mouthrinse (essential oil-containing mouthrinse) once a day after brushing for up to 4 Weeks.
Arm/Group | Negative Control Group (Toothbrushing Only) | Device Control Group (Toothbrushing, Device + Water) | Test Group (Toothbrushing, Device + Oil-containing Mouthrinse)
Number analyzed (Participants) | 42 | 44 | 44
Units on a scale | 2.674 (0.0432) | 2.213 (0.0422) | 2.005 (0.0422)
Statistical Analysis 1: Comparison: Negative Control Group (Toothbrushing Only) vs Device Control Group (Toothbrushing, Device + Water); Statistical analysis at Week 4; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.461, 95% CI 2-sided [-0.581 to -0.341]
Statistical Analysis 2: Comparison: Negative Control Group (Toothbrushing Only) vs Test Group (Toothbrushing, Device + Oil-containing Mouthrinse); Statistical analysis at Week 4; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.669, 95% CI 2-sided [-0.789 to -0.549]
Statistical Analysis 3: Comparison: Device Control Group (Toothbrushing, Device + Water) vs Test Group (Toothbrushing, Device + Oil-containing Mouthrinse); Test type: Superiority — Statistical analysis at Week 4; p < 0.001, ANCOVA; Difference in LS mean = -0.208, 95% CI 2-sided [-0.326 to -0.090]

2. Primary Outcome: Whole-mouth Mean Plaque Index at Week 4
Description: Plaque area was scored using the Turesky modification of the Quigley-Hein Plaque Index (PI), on six surfaces (distobuccal, midbuccal and mesiobuccal, distolingual, midlingual and mesiolingual) of all scorable teeth, using following score range; 0: indicates no plaque; 1: separate flecks or discontinuous band of plaque on the gingival (cervical) margin; 2: thin (up to 1 mm), continuous band of plaque at the gingival margin; 3: band of plaque wider than 1mm but less than1/3 of the surface; 4: plaque covering 1/3 or more, but less than 2/3 of the surface; 5 plaque covering 2/3 or more of the surface.
Time Frame: Week 4
Population: FAS included all randomized participants who used study product and had baseline and at least one data for mean PI post baseline.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Negative Control Group (Toothbrushing Only) | Device Control Group (Toothbrushing, Device + Water) | Test Group (Toothbrushing, Device + Oil-containing Mouthrinse)
Number analyzed (Participants) | 42 | 44 | 44
Units on a scale | 2.545 (0.0473) | 2.051 (0.0462) | 1.848 (0.0462)
Statistical Analysis 1: Comparison: Negative Control Group (Toothbrushing Only) vs Device Control Group (Toothbrushing, Device + Water); Statistical analysis at Week 4; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.494, 95% CI 2-sided [-0.625 to -0.363]
Statistical Analysis 2: Comparison: Negative Control Group (Toothbrushing Only) vs Test Group (Toothbrushing, Device + Oil-containing Mouthrinse); Statistical analysis at Week 4; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.697, 95% CI 2-sided [-0.828 to -0.567]
Statistical Analysis 3: Comparison: Device Control Group (Toothbrushing, Device + Water) vs Test Group (Toothbrushing, Device + Oil-containing Mouthrinse); Statistical analysis at Week 4; Test type: Superiority; p = 0.002, ANCOVA; Difference in LS mean = -0.203, 95% CI [-0.333 to -0.074]

3. Secondary Outcome: Interproximal Mean Modified Gingival Index (Mean MGI) at Week 2 and 4
Description: Gingivitis was assessed by the MGI on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth as per following score range: 0 indicates normal (absence of inflammation;) 1 indicates mild inflammation (slight change in color, little change in texture) of any portion of the entire gingival unit; 2 indicates mild inflammation of the entire gingival unit; 3 indicates moderate inflammation (moderate glazing, redness, edema, and/or hypertrophy) of the gingival unit. 4 indicates severe inflammation (marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration) of the gingival unit.
Time Frame: Week 2 and 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Negative Control Group (Toothbrushing Only) | Device Control Group (Toothbrushing, Device + Water) | Test Group (Toothbrushing, Device + Oil-containing Mouthrinse)
Number analyzed (Participants) | 42 | 44 | 44
Units on a scale
  Week 2 | 2.067 (0.0069) | 2.027 (0.0067) | 2.023 (0.0068)
  Week 4 | 2.071 (0.0108) | 1.980 (0.0106) | 1.927 (0.0107)
Statistical Analysis 1: Comparison: Negative Control Group (Toothbrushing Only) vs Device Control Group (Toothbrushing, Device + Water); Statistical analysis at Week 2; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.040, 95% CI 2-sided [-0.059 to -0.021]
Statistical Analysis 2: Comparison: Negative Control Group (Toothbrushing Only) vs Test Group (Toothbrushing, Device + Oil-containing Mouthrinse); Statistical analysis at Week 2; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.044, 95% CI [-0.064 to -0.025]
Statistical Analysis 3: Comparison: Device Control Group (Toothbrushing, Device + Water) vs Test Group (Toothbrushing, Device + Oil-containing Mouthrinse); Statistical analysis at Week 2; Test type: Superiority; p = 0.671, ANCOVA; Difference in LS mean = -0.004, 95% CI 2-sided [-0.023 to 0.015]
Statistical Analysis 4: Comparison: Negative Control Group (Toothbrushing Only) vs Device Control Group (Toothbrushing, Device + Water); Statistical analysis at Week 4; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.091, 95% CI 2-sided [-0.121 to -0.061]
Statistical Analysis 5: Comparison: Negative Control Group (Toothbrushing Only) vs Test Group (Toothbrushing, Device + Oil-containing Mouthrinse); Statistical analysis at Week 4; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.144, 95% CI 2-sided [-0.175 to -0.114]
Statistical Analysis 6: Comparison: Device Control Group (Toothbrushing, Device + Water) vs Test Group (Toothbrushing, Device + Oil-containing Mouthrinse); Statistical analysis at Week 4; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.053, 95% CI 2-sided [-0.083 to -0.023]

4. Secondary Outcome: Whole-mouth Modified Gingival Index (Mean MGI) at Week 2 and 4
Description: as for outcome 3
Time Frame: Week 2 and 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Negative Control Group (Toothbrushing Only) | Device Control Group (Toothbrushing, Device + Water) | Test Group (Toothbrushing, Device + Oil-containing Mouthrinse)
Number analyzed (Participants) | 42 | 44 | 44
Units on a scale
  Week 2 | 2.142 (0.0091) | 2.052 (0.0089) | 1.979 (0.0090)
  Week 4 | 2.144 (0.0109) | 1.995 (0.0106) | 1.888 (0.0107)
Statistical Analysis 1: Comparison: Negative Control Group (Toothbrushing Only) vs Device Control Group (Toothbrushing, Device + Water); Statistical analysis at Week 2; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.090, 95% CI 2-sided [-0.115 to -0.065]
Statistical Analysis 2: Comparison: Negative Control Group (Toothbrushing Only) vs Test Group (Toothbrushing, Device + Oil-containing Mouthrinse); Statistical analysis at Week 2; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.164, 95% CI 2-sided [-0.189 to -0.138]
Statistical Analysis 3: Comparison: Device Control Group (Toothbrushing, Device + Water) vs Test Group (Toothbrushing, Device + Oil-containing Mouthrinse); Statistical analysis at Week 2; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.073, 95% CI 2-sided [-0.099 to -0.048]
Statistical Analysis 4: Comparison: Negative Control Group (Toothbrushing Only) vs Device Control Group (Toothbrushing, Device + Water); Statistical analysis at Week 4; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.150, 95% CI 2-sided [-0.180 to -0.120]
Statistical Analysis 5: Comparison: Negative Control Group (Toothbrushing Only) vs Test Group (Toothbrushing, Device + Oil-containing Mouthrinse); Statistical analysis at Week 4; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.257, 95% CI 2-sided [-0.287 to -0.226]
Statistical Analysis 6: Comparison: Device Control Group (Toothbrushing, Device + Water) vs Test Group (Toothbrushing, Device + Oil-containing Mouthrinse); Statistical analysis at Week 4; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.107, 95% CI 2-sided [-0.137 to -0.077]

5. Secondary Outcome: Interproximal Mean Plaque Index (Mean PI) at Week 2
Description: as for outcome 2
Time Frame: Week 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Negative Control Group (Toothbrushing Only) | Device Control Group (Toothbrushing, Device + Water) | Test Group (Toothbrushing, Device + Oil-containing Mouthrinse)
Number analyzed (Participants) | 42 | 44 | 44
Units on a scale | 2.794 (0.0372) | 2.431 (0.0364) | 2.260 (0.0364)
Statistical Analysis 1: Comparison: Negative Control Group (Toothbrushing Only) vs Device Control Group (Toothbrushing, Device + Water); Statistical analysis at Week 2; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.362, 95% CI 2-sided [-0.465 to -0.259]
Statistical Analysis 2: Comparison: Negative Control Group (Toothbrushing Only) vs Test Group (Toothbrushing, Device + Oil-containing Mouthrinse); Statistical analysis at Week 2; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.534, 95% CI 2-sided [-0.637 to -0.431]
Statistical Analysis 3: Comparison: Device Control Group (Toothbrushing, Device + Water) vs Test Group (Toothbrushing, Device + Oil-containing Mouthrinse); Statistical analysis at Week 2; Test type: Superiority; p = 0.001, ANCOVA; Difference in LS mean = -0.171, 95% CI 2-sided [-0.273 to -0.069]

6. Secondary Outcome: Whole-mouth Mean Plaque Index (Mean PI) at Week 2
Description: as for outcome 2
Time Frame: Week 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Negative Control Group (Toothbrushing Only) | Device Control Group (Toothbrushing, Device + Water) | Test Group (Toothbrushing, Device + Oil-containing Mouthrinse)
Number analyzed (Participants) | 42 | 44 | 44
Units on a scale | 2.688 (0.0395) | 2.287 (0.0386) | 2.130 (0.0386)
Statistical Analysis 1: Comparison: Negative Control Group (Toothbrushing Only) vs Device Control Group (Toothbrushing, Device + Water); Statistical analysis at Week 2; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.401, 95% CI 2-sided [-0.510 to -0.292]
Statistical Analysis 2: Comparison: Negative Control Group (Toothbrushing Only) vs Test Group (Toothbrushing, Device + Oil-containing Mouthrinse); Statistical analysis at Week 2; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.558, 95% CI 2-sided [-0.667 to -0.449]
Statistical Analysis 3: Comparison: Device Control Group (Toothbrushing, Device + Water) vs Test Group (Toothbrushing, Device + Oil-containing Mouthrinse); Statistical analysis at Week 2; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.157, 95% CI 2-sided [-0.265 to -0.049]

7. Secondary Outcome: Interproximal Mean Bleeding Index (Mean BI) at Week 2 and 4
Description: Bleeding was assessed using the Gingival BI. A periodontal probe with a 0.5 millimeter (mm) diameter tip was inserted into the gingival crevice, and swept from distal to mesial around the tooth at an angle of approximately 60 degree, while in contact with the sulcular epithelium. Each of four gingival areas (distobuccal, midbuccal, mid-lingual, and mesiolingual) around each tooth was assessed. After approximately 30 seconds, bleeding at each gingival unit was recorded according to the following scale: 0 indicates absence of bleeding after 30 seconds; 1 indicates bleeding after 30 seconds; 2 indicates immediate bleeding.
Time Frame: Week 2 and 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Negative Control Group (Toothbrushing Only) | Device Control Group (Toothbrushing, Device + Water) | Test Group (Toothbrushing, Device + Oil-containing Mouthrinse)
Number analyzed (Participants) | 42 | 44 | 44
Units on a scale
  Week 2 | 0.059 (0.0058) | 0.028 (0.0057) | 0.020 (0.0057)
  Week 4 | 0.052 (0.0059) | 0.033 (0.0057) | 0.018 (0.0058)
Statistical Analysis 1: Comparison: Negative Control Group (Toothbrushing Only) vs Device Control Group (Toothbrushing, Device + Water); Statistical analysis at Week 2; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.030, 95% CI 2-sided [-0.046 to -0.014]
Statistical Analysis 2: Comparison: Negative Control Group (Toothbrushing Only) vs Test Group (Toothbrushing, Device + Oil-containing Mouthrinse); Statistical analysis at Week 2; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.039, 95% CI 2-sided [-0.055 to -0.023]
Statistical Analysis 3: Comparison: Device Control Group (Toothbrushing, Device + Water) vs Test Group (Toothbrushing, Device + Oil-containing Mouthrinse); Statistical analysis at Week 2; Test type: Superiority; p = 0.294, ANCOVA; Difference in LS mean = -0.009, 95% CI 2-sided [-0.025 to 0.007]
Statistical Analysis 4: Comparison: Negative Control Group (Toothbrushing Only) vs Device Control Group (Toothbrushing, Device + Water); Statistical analysis at Week 4; Test type: Superiority; p = 0.020, ANCOVA; Difference in LS mean = -0.019, 95% CI 2-sided [-0.035 to -0.003]
Statistical Analysis 5: Comparison: Negative Control Group (Toothbrushing Only) vs Test Group (Toothbrushing, Device + Oil-containing Mouthrinse); Statistical analysis at Week 4; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.034, 95% CI 2-sided [-0.050 to -0.018]
Statistical Analysis 6: Comparison: Device Control Group (Toothbrushing, Device + Water) vs Test Group (Toothbrushing, Device + Oil-containing Mouthrinse); Statistical analysis at Week 4; Test type: Superiority; p = 0.071, ANCOVA; Difference in LS mean = -0.015, 95% CI 2-sided [-0.031 to 0.001]

8. Secondary Outcome: Whole-mouth Mean Bleeding Index (Mean BI) at Week 2 and 4
Description: as for outcome 7
Time Frame: Week 2 and 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Negative Control Group (Toothbrushing Only) | Device Control Group (Toothbrushing, Device + Water) | Test Group (Toothbrushing, Device + Oil-containing Mouthrinse)
Number analyzed (Participants) | 42 | 44 | 44
Units on a scale
  Week 2 | 0.160 (0.0059) | 0.094 (0.0058) | 0.078 (0.0058)
  Week 4 | 0.154 (0.0065) | 0.077 (0.0064) | 0.052 (0.0064)
Statistical Analysis 1: Comparison: Negative Control Group (Toothbrushing Only) vs Device Control Group (Toothbrushing, Device + Water); Statistical analysis at Week 2; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.067, 95% CI [-0.083 to -0.050]
Statistical Analysis 2: Comparison: Negative Control Group (Toothbrushing Only) vs Test Group (Toothbrushing, Device + Oil-containing Mouthrinse); Statistical analysis at Week 2; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.083, 95% CI 2-sided [-0.099 to -0.066]
Statistical Analysis 3: Comparison: Device Control Group (Toothbrushing, Device + Water) vs Test Group (Toothbrushing, Device + Oil-containing Mouthrinse); Statistical analysis at Week 2; Test type: Superiority; p = 0.057, ANCOVA; Difference in LS mean = -0.016, 95% CI 2-sided [-0.032 to 0.000]
Statistical Analysis 4: Comparison: Negative Control Group (Toothbrushing Only) vs Device Control Group (Toothbrushing, Device + Water); Statistical analysis at Week 4; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.077, 95% CI 2-sided [-0.095 to -0.059]
Statistical Analysis 5: Comparison: Negative Control Group (Toothbrushing Only) vs Test Group (Toothbrushing, Device + Oil-containing Mouthrinse); Statistical analysis at Week 4; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -0.101, 95% CI 2-sided [-0.120 to -0.083]
Statistical Analysis 6: Comparison: Device Control Group (Toothbrushing, Device + Water) vs Test Group (Toothbrushing, Device + Oil-containing Mouthrinse); Statistical analysis at Week 4; Test type: Superiority; p = 0.009, ANCOVA; Difference in LS mean = -0.024, 95% CI 2-sided [-0.042 to -0.006]

ADVERSE EVENTS:
Time Frame: Up to 4 Weeks
Description: Safety analysis set consisted of all randomized participants who used study product.
Arm/Group | Negative Control Group (Toothbrushing Only) | Device Control Group (Toothbrushing, Device + Water) | Test Group (Toothbrushing, Device+ Oil-containing Mouthrinse)
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/47 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 0/46 | 0/47 | 0/47

LIMITATIONS AND CAVEATS:
No study limitation was reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.